CLINICAL TRIAL: NCT06614088
Title: Serum Calprotectin in Surgical Septic Patients as an Early Predictor of Clinical Severity and Mortality: a Prospective Comparative Study.
Brief Title: Serum Calprotectin in Surgical Septic Patients
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Dario Tartaglia, dr, Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: 11 2021
Record Dates: First submitted 2023-08-11; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Infection, Intraabdominal; Sepsis Abdominal; Biomarker
Keywords: Serum calprotectin; Surgical infections
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Eligible patients with CPIRO 0-2
  Interventions: Diagnostic Test: serum calprotectin
- Group B: Eligible patients with CPIRO >3
  Interventions: Diagnostic Test: serum calprotectin
- Group C: Control group (elective surgical patients without any source of intra-abdominal infection)
  Interventions: Diagnostic Test: serum calprotectin

INTERVENTIONS:
Diagnostic Test: serum calprotectin — A blood sample is collected at time of admission to detect serum level of calprotectin

SUMMARY:
To early evaluate the serum levels of calprotectin in patients suffering from intra-abdominal sepsis requiring a surgical treatment. The research project aims to investigate the role of serum calprotectin in the diagnosis of sepsis and to establish whether its level significantly correlates with different degree of disease severity and with short and long-term outcomes. If these associations were confirmed, serum calprotectin would represent an easily and rapidly detectable biomarker able to predict the severity of sepsis.

DETAILED DESCRIPTION:
Inclusion criteria are age>18 years; diagnosis of upper/lower gastro-intestinal perforation, intestinal occlusion, acute cholecystitis, acute appendicitis or intra-abdominal sepsis.

Enrolled patients will be divided in two groups according to the Calgary PIRO (CPIRO) score evaluation: group A includes patients with CPIRO score </= 2 and represents patient with mild form of intra-abdominal sepsis while group B includes patients with CPIRO score >/= 3, therefore representing patients with more severe systemic forms. The control group (group C) will be made by elective surgical adult patients.

A blood sample will be collected in sample tubes without anticoagulant from all the eligible patients at admission. After centrifugation, the serum will be stored at -80°C until analysis. The serum level of calprotectin will be measured using a commercially available ELISA Kit based on polyclonal antibodies, according to the manufacturer instruction and fully blinded to any clinical data of the patients or controls.

To our knowledge, this is going to be the first study comparing the levels of serum calprotectin in a large cohort of surgical patients with different degree of intra-abdominal sepsis.

Our primary outcome is to determine whether the serum calprotectin level at the admission is increased in septic patients compared to the control group. We will correlate serum calprotectin level with PCT levels, to check which is the most accurate for the detection of sepsis. Our secondary outcome is to analyze if serum calprotectin level at admission correlates with the clinical severity of sepsis, evaluated trough the CPIRO score. Finally, we will verify if calprotectin level at admission is predictive of short and long-term morbidity and mortality, need for ICU admission and invasive/non-invasive post-operative reinterventions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of upper/lower gastro-intestinal perforation
* diagnosis of intestinal occlusion
* diagnosis of acute cholecystitis
* diagnosis of complicated acute appendicitis
* radiological diagnosis of intra-abdominal sepsis

Exclusion Criteria:

* recent (<3 months) surgery
* recent (<3 months) trauma
* diagnosis of acute pancreatitis
* diagnosis of burn

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Septic patients requiring surgery at the Department of General and Emergency Surgery of the University of Pisa
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Sepsis detection | admission
  We'll measure the serum calprotectin level in enrolled patients of the two groups (group A and B) and in patients of the control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Pisana (AOUP), Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Simm M, Soderberg E, Larsson A, Castegren M, Nilsen T, Eriksson M, Lipcsey M. Performance of plasma calprotectin as a biomarker of early sepsis: a pilot study. Biomark Med. 2016 Aug;10(8):811-8. doi: 10.2217/bmm-2016-0032. Epub 2016 Jul 14. PMID 27414210
- [Background] Larsson A, Tyden J, Johansson J, Lipcsey M, Bergquist M, Kultima K, Mandic-Havelka A. Calprotectin is superior to procalcitonin as a sepsis marker and predictor of 30-day mortality in intensive care patients. Scand J Clin Lab Invest. 2020 Feb-Apr;80(2):156-161. doi: 10.1080/00365513.2019.1703216. Epub 2019 Dec 14. PMID 31841042